CLINICAL TRIAL: NCT00638599
Title: Comparison of Laryngeal Mask Airway (LMA®) and Tracheal Tube for Airway Management in Modified Radical Mastectomy on Breast Cancer
Brief Title: Comparison of Laryngeal Mask Airway (LMA®) and Tracheal Tube in Modified Radical Mastectomy on Breast Cancer
Acronym: LMATBBC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: XiRong Guo, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NMU-2579-7FW; NMU075451
Record Dates: First submitted 2008-03-04; First posted 2008-03-19 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2009-07

CONDITIONS: Breast Cancer
Keywords: Intubation, intratracheal; Homeostasis; Mastectomy, modified radical; Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): LMA® is placed after anesthesia induction till the end of operation
  Interventions: Device: LMA®
- 2 (Active Comparator): Standard tracheal tube is inserted after anesthesia induction till the end of operation
  Interventions: Device: Endotracheal tube

INTERVENTIONS:
Device: LMA® — LMA® is placed after anesthesia induction and removed after the operation
  Arms: 1
Device: Endotracheal tube — Standard endotracheal tube is inserted after anesthesia induction and extubated after the operation
  Arms: 2

SUMMARY:
Airway management in anesthesia is critical to guarantee appropriate treatment of possible respiratory complications and successful operative practice. LMA® is an alternative to tracheal tube in some surgeries like as mastectomy on breast cancer. Given no need using muscular relaxants in mastectomy, the investigators hypothesized that LMA® would be a superior manner in airway management in radical modified mastectomy on breast cancer than the tracheal tube, and the LMA® might produce less influence on patients' circulatory homeostasis, and easier to be placed before operation.

ELIGIBILITY:
Inclusion Criteria:

* Chinese
* Diagnosed breast cancer
* Undergoing modified radical mastectomy
* Agreed to participate the study with informed contract.

Exclusion Criteria:

* Organic dysfunction
* Long-lasting post-anesthetic care unit(PACU) staying.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Circulatory Homeostasis | 15min prior to operation to 15min posterior to operation

SECONDARY OUTCOMES:
Airway pressure | 15min prior to operation to 15min posterior to operation
Blood gas | 15min prior to operation to 15min posterior to operation
Airway complications | Start of operation to 6h after operation

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Director — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Health Care Hospital, Nanjing, Jiangsu, China